CLINICAL TRIAL: NCT04088487
Title: New in Town-Internet Intervention for Migrants: a Randomized Controlled Trial
Brief Title: New in Town-Internet Intervention for Migrants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention includes tasks that encourage participants to interact with the social environment which is unethical due to the outbreak of COVID-19.
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WP/2018/A/10
Record Dates: First submitted 2019-08-06; First posted 2019-09-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Self Efficacy; Loneliness; Social Skills
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants gain access to the internet intervention after the baseline measurement (pre-test).
  Interventions: Behavioral: New in Town-Interner Intervention for Migrants
- Waitlist control group (Other): Participants gain access to the internet intervention 8 weeks after the baseline measurement (pre-test).
  Interventions: Behavioral: New in Town-Interner Intervention for Migrants

INTERVENTIONS:
Behavioral: New in Town-Interner Intervention for Migrants — New in Town is an internet intervention for migrants that aims at increasing social self-efficacy. Exercises in the intervention are based on the principles of Cognitive Behavioral Therapy and relate to four sources of self-efficacy beliefs-mastery experiences, vicarious experiences, verbal persuasions, and emotional and physiological states (Bandura, 1997).

SUMMARY:
New in Town is an internet intervention for migrants that aims at increasing social self-efficacy. The study aim is to evaluate its effectiveness.

DETAILED DESCRIPTION:
The number of migrants worldwide is growing rapidly over the past years. Migration often requires creating a whole new social network. There is something that can help migrants to do it-their beliefs. Social self-efficacy is confidence in ability to engage in social interactional tasks necessary to initiate and maintain interpersonal relationships. These beliefs are positively related to social adjustment and negatively related to acculturative stress, depression, and loneliness. Therefore, social self-efficacy may be potentially beneficial for the psychological adjustment of migrants helping them establish new connections in the social environment. Based on this observation the investigators have created New in Town, an internet intervention. Exercises in the intervention are based on the principles of Cognitive Behavioral Therapy and relate to four sources of self-efficacy beliefs-mastery experiences, vicarious experiences, verbal persuasions, and emotional and physiological states.

The effectiveness of New in Town intervention will be tested in a two-arm randomized controlled trial with waitlist control group. Primary outcome is social self-efficacy, and secondary outcomes include loneliness, perceived social support, and satisfaction with life. Other measure of interest is system usability. Participants will be assessed at pre-test (T1), 3-week post-tests (T2), as well as 8-week follow-up (T3). The investigators aim to analyze the effect size of the intervention and between-groups comparisons at post-test and follow-up.

This study will provide insights into the effectiveness of an internet intervention in increasing social self-efficacy, perceived social support and satisfaction with life, and reducing loneliness.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* having changed the place of residence in the last 6 months

Exclusion Criteria:

- no access to a internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Change on Social Self-Efficacy | Change from baseline on Social Self-Efficacy (3 weeks)
  Social self-efficacy will be measured with the General Self-efficacy Scale (GSES). The measure consists of two subscales for measuring 1) generalized beliefs about self-efficacy (17 test items) and 2) beliefs about self-efficacy in establishing and maintaining relationships with others (6 test items). The remaining test items (7) are buffer theorems. The respondents give answers on a scale 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). In the trial, the investigators will use one subscale, which is beliefs about self-efficacy in establishing and maintaining relationships with others. Social self-efficacy will be indicated by the total sum of 6 items scores. The higher total score represents higher social self-efficacy.
Change on Social Self-Efficacy | Change from baseline on Social Self-Efficacy (8 weeks)
  Social self-efficacy will be measured with the General Self-efficacy Scale (GSES). The measure consists of two subscales for measuring 1) generalized beliefs about self-efficacy (17 test items) and 2) beliefs about self-efficacy in establishing and maintaining relationships with others (6 test items). The remaining test items (7) are buffer theorems. The respondents give answers on a scale 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). In the trial, the investigators will use one subscale, which is beliefs about self-efficacy in establishing and maintaining relationships with others. Social self-efficacy will be indicated by the total sum of 6 items scores. The higher total score represents higher social self-efficacy.

SECONDARY OUTCOMES:
Change on Loneliness | Change from baseline on Loneliness (3 weeks)
  To measure loneliness, the investigators will use De Jong Gierveld Loneliness Scale. The scale is composed of 11 items; 6 of them are formulated negatively and 5 positively. Each item is measured using on 5-point Likert scale (1 = definitely yes, 5 = definitely no). Positive items should be reversed. The sum of scores is counted on 2 separate subscales: emotional and social loneliness. The higher total score represents higher loneliness.
Change on Loneliness | Change from baseline on Loneliness (8 weeks)
  To measure loneliness, the investigators will use De Jong Gierveld Loneliness Scale. The scale is composed of 11 items; 6 of them are formulated negatively and 5 positively. Each item is measured using on 5-point Likert scale (1 = definitely yes, 5 = definitely no). Positive items should be reversed. The sum of scores is counted on 2 separate subscales: emotional and social loneliness. The higher total score represents higher loneliness.
Change on Social support | Change from baseline on Social support (3 weeks)
  To measure social support, the investigators will use The Berlin Social Support Scale (BSSS). The scale consists of 6 subscales: perceived available support, need for support, support seeking, actually received support (recipient), provided support (provider), protective buffering scale. The BSSS contains 32 items that are scored on a 4-point scale (1 = strongly disagree, 4 = strongly agree). Before scoring items negative ones need to be reversed. Scores will be counted both on a general scale and subscales. In the trial, only 3 of 6 subscales will be applied: perceived available support (8 test items), need for support (4 test items), and support seeking (5 test items). The higher total score represents higher social support.
Change on Social support | Change from baseline on Social support (8 weeks)
  To measure social support, the investigators will use The Berlin Social Support Scale (BSSS). The scale consists of 6 subscales: perceived available support, need for support, support seeking, actually received support (recipient), provided support (provider), protective buffering scale. The BSSS contains 32 items that are scored on a 4-point scale (1 = strongly disagree, 4 = strongly agree). Before scoring items negative ones need to be reversed. Scores will be counted both on a general scale and subscales. In the trial, only 3 of 6 subscales will be applied: perceived available support (8 test items), need for support (4 test items), and support seeking (5 test items). The higher total score represents higher social support.
Change on Satisfaction with life | Change from baseline on Satisfaction with life (3 weeks)
  To measure satisfaction with life, the investigators will use The Satisfaction with Life Scale (SWLS). It is a short scale to assess perceived satisfaction with one's life. It consists of 5 items. The respondents provide answers on a 7-point scale (1 = strongly disagree, 7 = strongly agree). Possible scores range from 5 to 35, while score of 20 indicates a neutral point. The higher total score represents higher satisfaction with life.
Change on Satisfaction with life | Change from baseline on Satisfaction with life (8 weeks)
  To measure satisfaction with life, the investigators will use The Satisfaction with Life Scale (SWLS). It is a short scale to assess perceived satisfaction with one's life. It consists of 5 items. The respondents provide answers on a 7-point scale (1 = strongly disagree, 7 = strongly agree). Possible scores range from 5 to 35, while score of 20 indicates a neutral point. The higher total score represents higher satisfaction with life.

OTHER OUTCOMES:
System usability | 3-week post-test (only experimental group)
  An overall impression of the intervention will be assessed by The User Experience Questionnaire (UEQ). It is a self-reported measure that contains 6 subscales: attractiveness, perspicuity, efficiency, dependability, stimulation, novelty. Participants respond to 26 items using a 7-point scale (-3 = the most negative answer, 0 = neutral, +3 = the most positive answer). User experience will only be assessed at post-test among participants allocated to the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rogala, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities
Locations (1):
- SWPS University of Social Sciences and Humanities, Warsaw, Warszawa, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandura, A. (1997). Self-efficacy: The exercise of control. Macmillan.
- [Background] Connolly, J. (1989). Social self-efficacy in adolescence: Relations with self-concept, social adjustment, and mental health. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement, 21(3), 258.
- [Background] Constantine MG, Okazaki S, Utsey SO. Self-concealment, social self-efficacy, acculturative stress, and depression in African, Asian, and Latin American international college students. Am J Orthopsychiatry. 2004 Jul;74(3):230-241. doi: 10.1037/0002-9432.74.3.230. PMID 15291700
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Gierveld, J. D. J., & Van Tilburg, T. (1999). Manual of the loneliness scale. Amsterdam: Department of Social Research Methodology.
- [Background] Łuszczyńska, A., Mazurkiewicz, M., Kowalska, M., & Schwarzer, R. (2006). Berlińskie skale wsparcia społecznego (BSSS): Wyniki wstępnych badań nad adaptacją skal i ich własnośnciami psychometrycznymi = Berlin social support scales (BSSS): Polish version of BSSS and preliminary results on its psychometric properties. Studia Psychologiczne, 44(3), 17-27.
- [Background] Sherer, M., Maddux, J. E., Mercandante, B., Prentice-Dunn, S., Jacobs, B., & Rogers, R. W. (1982). The self-efficacy scale: Construction and validation. Psychological reports, 51(2), 663-671.
- [Background] Smith, H. M., & Betz, N. E. (2000). Development and validation of a scale of perceived social self-efficacy. Journal of Career Assessment, 8(3), 283-301.
- [Background] Schrepp, M., Pérez Cota, M., Gonçalves, R., Hinderks, A., & Thomaschewski, J. (2017). Adaption of user experience questionnaires for different user groups. Universal Access in the Information Society, 16(3), 629-640.
- [Background] United Nations (2017). 2017 International Migration Report.
- [Derived] Maj A, Matynia M, Michalak N, Bis A, Andersson G. New in Town-An internet-based self-efficacy intervention for internal migrants: A randomized controlled trial. PLoS One. 2024 Mar 7;19(3):e0299638. doi: 10.1371/journal.pone.0299638. eCollection 2024. PMID 38452136
- [Derived] Rogala A, Szczepaniak M, Michalak N, Andersson G. Internet-based self-help intervention aimed at increasing social self-efficacy among internal migrants in Poland: Study protocol for a randomized controlled trial. Internet Interv. 2020 Apr 23;21:100322. doi: 10.1016/j.invent.2020.100322. eCollection 2020 Sep. PMID 32328440